CLINICAL TRIAL: NCT03596996
Title: Optimizing Iron Status While Minimizing Morbidity in HIV-infected Ugandan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Joint Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1608M92324
Record Dates: First submitted 2018-06-05; First posted 2018-07-24 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Anemia; Iron-deficiency; Iron Deficiency Anemia; Hiv
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Acquired Immunodeficiency Syndrome | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous Sulfate (Experimental): Children 6 to 23 months of age will receive a tablet that contains the equivalent of 12.5 mg of elemental iron. Children over 24 months will receive a tablet that contains the equivalent of 30 mg of elemental iron.
  Interventions: Dietary Supplement: Ferrous Sulfate
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate — Ferrous sulfate dosed by WHO guidelines by age for the prevention of iron deficiency and anemia.
  Arms: Ferrous Sulfate
Dietary Supplement: Placebo — Placebo with identical appearance comparison intervention arm
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled trial of the effect of 84 days of daily iron supplementation on iron status, gut microbiome profile, infectious disease frequency, and HIV disease severity in moderately anemic [hemoglobin 9 - <11 g/dL (6-59 mo); hemoglobin 9 - < 11.5 g/dL (5 -12 years)], HIV-infected Ugandan children between the ages of 6 mos and 12 years.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of HIV (based JCRC clinic records);
2. On Highly Active Antiretroviral Treatment (HAART) for ≥ 6 months
3. Age 6 months - 12 years at the time of screening
4. Hemoglobin 9 - <11 g/dL (6-59 mo); hemoglobin 9 - < 11.5 g/dL (5 -12 years)by CBC at time of screening

Exclusion Criteria:

1. Acute illness or current opportunistic infection
2. Temperature >= 38.0°C at the time of screening
3. Known sickle cell disease
4. Acute malnutrition (bilateral pitting edema or extreme wasting)
5. Any chronic illness requiring regular medical attention
6. Residence > 50 km from JCRC hospital
7. Non-English or Luganda speaking
8. Currently taking iron supplements

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 3 months
  Measurement of hemoglobin
Anemia | 3 months
  Prevalence of anemia
Iron status | 3 months
  Iron status measured using ferritin, sTfR, CRP and hepcidin concentration in plasma

SECONDARY OUTCOMES:
Sick Child Visits | 3 months
  Number of acute illnesses leading to visit to healthcare provider
Dietary iron absorption | 2 weeks
  Percentage of 57Fe from oral dose that is incorporated into hemoglobin
HIV virologic control | 3 month
  HIV viral load
HIV related immunosuppression | 3 months
  CD4 count

OTHER OUTCOMES:
Microbiome gut profile | 3 months
  Ratio of Enterobacteriaceae to Lactobacillaceae and Bifidobacteriaceae

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cusick, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Joint Clinical Research Centre, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD used for the current study are available after publication of primary findings on reasonable request. Requests may be subject to review by Joint Clinical Research Centre in Kampala, Uganda to determine if aims and analysis are consistent with participant consent.
Access Criteria: Joint Clinical Research Centre review to determine if aims and analysis on consistent with participant consent.

REFERENCES:
- [Derived] Frosch AEP, Musiime V, Staley C, Conroy AL, Rutebarika D, Ategeka G, Cusick SE. Safety and efficacy of iron supplementation with 3 months of daily ferrous sulphate in children living with HIV and mild-to-moderate anaemia in Uganda: a double-blind, randomised, placebo-controlled trial. Lancet HIV. 2024 Nov;11(11):e727-e735. doi: 10.1016/S2352-3018(24)00238-8. Epub 2024 Oct 11. PMID 39401504